CLINICAL TRIAL: NCT00146874
Title: Cardiac Resynchronization Therapy Registry Evaluating Patient Response With RENEWAL Family Devices
Brief Title: CRT RENEWAL Registry
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Other Study IDs: CR-CA-042704-H
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2006-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: cardiac resynchronization therapy

SUMMARY:
This registry will provide detailed patient demographics and characteristics at the time of enrollment and will also provide data regarding predictors of clinical outcomes such as heart failure decompensation, heart failure hospitalization, NYHA class, and quality of life.

DETAILED DESCRIPTION:
The CRT RENEWAL Registry aims to characterize patient demographics and clinical attributes at enrollment and overall event rates as defined by heart failure decompensation, heart failure hospitalization, death, and ventricular arrhythmic events. The registry will also assess clinical outcomes including quality of life (QOL), physical activity habits, and events rates, along with device diagnostics such as Activity Log Index and heart rate

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet current indications for the CONTAK RENEWAL® family of CRT-P or CRT-D devices
* Patients who receive either transvenous Guidant manufactured ventricular leads or non-Guidant epicardial leads
* Patients who have had an ejection fraction measured within six months of enrollment
* Patients who sign and date a Patient Informed Consent form at the enrollment visit
* Patients who remain in the clinical care of the enrolling physician in approved centers

Exclusion Criteria:

* Patients who are expected to receive a heart transplant during the duration of the registry
* Patients who currently have or who are likely to receive a tricuspid valve prosthesis
* Patients who are currently enrolled in another observational registry or investigational study that would directly impact the treatment or outcome of the CRT RENEWAL Registry. Each instance will be brought to the attention of Guidant's Clinical Application Research Studies (CARS) Department to determine eligibility
* Patients who are younger than 18 years of age
* Patients who are mentally incompetent and cannot sign a Patient Informed Consent form or comply with the registry
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Standard CRT population
Sampling Method: Non-Probability Sample
Enrollment: 1000
Dates: Start 2004-05; Primary Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kaplan, MD, Principal Investigator — Tri-City Cardiology Consultants